CLINICAL TRIAL: NCT03537391
Title: Imaging for Prostate Cancer Metastasis Detection - Traditional Imaging (Bone Scan and CT) Versus PSMA-PET-CT, SPECT-CT and Whole-Body MRI
Brief Title: Novel Imaging in Staging of Primary Prostate Cancer
Acronym: PROSTAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T95/2018
Record Dates: First submitted 2018-04-26; First posted 2018-05-25 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: High Risk Prostate Cancer
Keywords: prostate cancer; imaging of prostate cancer; staging of prostate cancer; prostate specific membrane antigen (PSMA); positron emission tomography; bone scintigraphy; whole body magnetic resonance imaging; whole body computer tomography; single photon emission tomography (SPECT)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: This is a prospective single-institutional study comparing the diagnostic accuracy of novel imaging modalities to traditional imaging modalities among high risk prostate cancer patients at initial diagnosis
Masking Description: Imaging modalities will be read blindly without the knowledge of results of the other imaging modalities. Readers will only know that a patient has prostate cancer with high risk for metastases. All imaging data will be analyzed visually with classifying lesions as normal, equivocal or metastatic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging based staging of high risk PC (Experimental): Each individual study patient will be imaged for PC metastasis detection with each different imaging modalities as follows:
  Traditional imaging (clinical standard imaging);
  1. Whole-body contrast enhanced computer tomography
  2. Planar bone scintigraphy
     Novel imaging (investigational imaging);
  3. SPECT/CT (investigational imaging)
  4. 18F-PSMA-PET/CT (investigational imaging)
  5. Whole-body MRI (investigational imaging)
  In order to define the true nature of the findings from each different imaging modality, comparison with best valuable comparator (BvC) is made. Consensus reading of all imaging modalities and follow-up data of clinical, imaging, histopathological and laboratory results are used to define BvC.
  Interventions: Diagnostic Test: Whole body contrast enhanced computer tomography; Diagnostic Test: 99mTC-HMDP planar bone scintigraphy (BS); Diagnostic Test: 99mTc-HMDP single photon emission computer tomography/computer tomography; Diagnostic Test: Whole-body magnetic resonance imaging; Diagnostic Test: Fluorine-18-prostate specific membrane antigen-1007- positron emission tomography/computer tomography

INTERVENTIONS:
Diagnostic Test: Whole body contrast enhanced computer tomography — Computed tomography of the thorax, abdomen and pelvis will be performed as a part of routine clinical evaluation protocol. The imaging will be done with contrast agent if there are no clinical contraindications for the use of contrast agent.
  Other Names: wbCE-CT
Diagnostic Test: 99mTC-HMDP planar bone scintigraphy (BS) — Planar bone scintigraphy will be performed as a part of routine clinical evaluation protocol. The subjects will be positioned supine on a Discovery NM/CT 670 CZT, a digital SPECT/CT scanner (General Electric Healthcare). The scanner includes a dual-detector, free-geometry integrated nuclear imaging camera with the advanced digital CZT detector technology combined with the high-performance Optima CT540 subsystem. Whole-body planar images will be scanned from the anterior and posterior views three hours after the intravenous injection of 670 MBq of 99mTc-HMDP. A wide-energy high-resolution (WEHR) collimator, a scan speed of 13 cm/min, a zoom of 1.0 and a matrix size of 256 x 1024 are used in the scintigraphy.
  Other Names: Planar BS
Diagnostic Test: 99mTc-HMDP single photon emission computer tomography/computer tomography — SPECT/CT imaging will be carried out after acquisition of the planar images with the same scanner. Three bed positions of SPECT data will be acquired from the top of the head to mid femoral level using WEHR collimators. A non-circular orbit, 60 views with 15-s scanning time per view will be acquired during 180 degrees of rotation. A 128 x 128 matrix size, a zoom of 1.0 and 15% photopeak and lower scatter energy windows are used. After SPECT a CT topogram and a low-dose tomogram with a modulated mAs (noise index ~ 70), 120 kVp, a pitch of 1.35 and a 2.5-mm slice thickness are scanned. The co-registration of SPECT and CT data is verified after which the SPECT images are reconstructed using modern iterative ordered subsets expectation (OSEM) reconstruction algorithm from General Electric or Hermes Medical Solutions, which includes, e.g., 10 iterations and 5 subsets and attenuation, collimator and scatter corrections.
  Other Names: SPECT/CT
Diagnostic Test: Whole-body magnetic resonance imaging — Magnetic resonance imaging examination will be performed using a 1.5T (Philips 1.5T Ingenia, Best, Netherlands and/or Siemens 1.5T Aera/Avant, Erlangen, Germany) or 3T (Philips 3T Ingenia, Best, Netherlands and/or Siemens 3T Skyra fit, Erlangen, German) MR system. The body matrix coil in combination with a spinal coil will be used for image acquisition. T1-weighted anatomic imaging, STIR fat suppressed images and DWI will be performed in axial and coronal directions. DWI will be obtained with single-shot 2D spin-echo echo-planar imaging. The total scan time will be approximately 50 minutes.
  Other Names: wbMRI
Diagnostic Test: Fluorine-18-prostate specific membrane antigen-1007- positron emission tomography/computer tomography — 18F-PSMA-1007 is produced by radiolabelling with fluorine-18 produced by irradiating oxygen-18. Administration of the formulated solution is done shortly (<10h) after production. Imaging is carried out with digital PET/CT scanner (Discovery MI;General Electric Medical Systems, Milwaukee, WI, USA). The patients receive intravenous injection of 200-300 MBq (3 MB/kg) of 18F-PSMA-1007 diluted in 3-5 ml of saline as a 60-sec bolus which will be promptly flushed with saline. Before data acquisition patients will be asked to void. A static emission scan will be acquired 60-min from tracer injection over whole body. The sinogram data will be corrected for deadtime, decay and photon attenuation and reconstructed in a 256x256 matrix. Image reconstruction follows a fully 3D maximum likelihood ordered subsets expectation maximization algorithm incorporating random and scatter correction with two iterations and 28 subsets.The final in-plane full-width half-maximum of the systems is < 6 mm.
  Other Names: 18F-PSMA-1007-PET/CT

SUMMARY:
Prostate cancer (PC) is the most common cancer among men and one quarter of diagnosed PC are metastatic at the time of diagnosis. Accurate staging is paramount as the stage is the most important factor when treatment decisions are made. The stage is also the single most important prognostic factor. Currently, traditional imaging methods for detection of PC metastasis, including bone scan (BS) and contrast enhanced whole-body computer tomography (CT), are rather inaccurate. Respectively, novel imaging techniques are evolving and novel imaging modalities are emerging in PC diagnostics and staging, but their clinical relevance is unclear and lacking prospective studies comparing traditional imaging with novel imaging.

This prospective single-institutional study compares the diagnostic accuracy of novel imaging modalities to traditional imaging modalities aiming to find the most appropriate staging modality in high-risk PC at the time of initial staging.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common cancer among men. The incidence of PC has increased dramatically in Finland since 1980´s and lately approximately 4.500 new PC cases have been diagnosed annually in Finland.

About one quarter of diagnosed PC are metastatic at the time of diagnosis. Accurate staging is extremely important, as the stage is single most important factor when treatment decisions are made and stage is the single most important prognostic factor. Localized PC is treated with active surveillance (low risk cases), or with treatment modalities with curative intent (radical prostatectomy or radiotherapy).Although recently radical treatments have been suggested to play a role in low volume metastatic disease, the standard treatment of metastatic disease is castration therapy.

In PC staging the most important anatomic locations to be imaged are i) bone, ii) lymph nodes (especially pelvic lymph nodes), and iii) extranodal soft tissues.

Detection of tumor bone metastases is commonly performed by BS. However, the results of recent studies have raised many doubts whether BS is as effective for confirming or excluding metastatic bone disease. Moreover, the sensitivity for 99mTc-methylene diphosphonate bone scintigraphy (99mTc-MDP BS) is only 50-70%. The detection of bone metastases in patients with high-risk PC is significantly improved by SPECT compared to planar BS. Other imaging modalities with potentially improved accuracy to detect bone metastases in PC include PET-scan and whole body MRI.

The value of positron emission tomography (PET) imaging depends on the suitability of used isotope tracer to identify lesions of the imaged tumor type. When bone is imaged with PET, 18F-fluoride has been the most commonly used tracer. Other commonly used PET tracers in PC include 18F-FDG, and 18F/11C-choline, but both have been late more or less replaced by PSMA-PET. Prostate-specific membrane antigen (PSMA) is a trans-membrane protein with an increased expression on cell membranes of PC cells. 68Ga-PSMA HBED-CC (Glu-NH-CO-NH-Lys- (Ahx)-[68Ga(HBED-CC)]) was designed as an extracellular PSMA inhibitor for PET imaging and has been shown to demonstrate high specificity for PSMA-expressing tumor cell. PSMA-PET results have been reported in several studies, but only in three prospective, one including 20-30 patients. Of those studies only study by Fendler and coworkers investigated overall staging, the other two studies by van Leeuwen focused on intraprostatic tumor detection or nodal metastases. Nevertheless, PSMA-PET/CT is a promising imaging modality both for soft tissues and bone. Recently 68Ga-PSMA was reported to outperform 99mTc-DPD-SPECT in detection of bone metastases in PC.

Recently, the novel PET tracer 18F-PSMA-1007 has been developed as a promising PSMA ligand to even outperform 68Ga-PSMA-PET in overall staging. 18F-PSMA-1007 have advantages in comparison to 68Ga-PSMA-PET including primary elimination of 18F-PSMA-1007 via the hepatobiliary excretion route leading to less isotope activity in urinary tract. Consequently, 18F-PSMA-1007 might lead to better local staging because of its favorable pharmacokinetics and tumor-specific uptake. 18F-PSMA-1007-PET combined with CT or even MRI could truly offer a 1-stop solution for both metastatic screening and local staging, but more prospective studies are needed to confirm this hypothesis.

Whole-body T1-weighted MRI is an effective method for bone imaging and is superior when compared to 99mTc-MDP BS. If combined with soft tissue imaging, bone and nodal imaging may be performed in single imaging session. Diffusion-weighted imaging (DWI) as a part of routine MRI examination is a promising tool for detection of an early intramedullary malignant lesion before cortical destruction or reactive processes due to bone marrow metastasis. DWI performs high contrast resolution between tumor and normal tissue. Individual variability of the mean apparent diffusion coefficient (ADC) values, as the result of DWI, may decrease the diagnostic accuracy of DWI. Diagnostic accuracy of DWI for detection of malignant lesion is better than 18-fluoro-deoxy-glucose (FDG) and for detection of bone metastasis is comparable to 11C-choline. However, it is unclear if it is superior compared to the standard T1-weighted imaging or STIR fat suppression technique. Currently there is not sufficient data comparing MRI and PSMA-PET/CT accuracy on bone imaging in PC.

In addition to bone, the possible tumor spread to soft tissues, especially pelvic lymph node is common in PC staging. Traditionally contrast enhanced abdomen and pelvic CT or MRI are used but the sensitivity of these imaging modalities is very limited. Diffusion-weighted MRI may improve the diagnostic accuracy when normal sized lymph nodes are evaluated. Still, different PET-tracers and recently especially 68Ga-PSMA and novel 18F-PSMA have both been considered as the most promising modalities for pelvic lymph node metastasis detection in PC and preliminary results suggest superior diagnostic accuracy of PSMA-PET compared to other modalities.

The investigators have previously investigated different imaging modalities for detection of bone metastases in prospective setting (Skeleta-trial). According to that study, 18F-NaF PET-CT and whole-body MRI are superior when compared to 99mTc-MDP SPECT-CT or 99mTc-MDP planar bone scan. Nevertheless, that study needs validation and further investigations as it was limited by low number (n=27) of PC patients, and PSMA-PET was not included in the study.

Clinicians face challenges when choosing optimal imaging modality/modalities for individual patient. Guidelines do not support any imaging in low risk cases. For some intermediate risk cases, and also for high-risk cases, if local treatment is planned, accurate staging of pelvic lymph node is important. In contrary, in very high-risk cases the knowledge of distant metastases is the single most important staging data. Optimally for clinicians most appropriate imaging technique would be chosen based on patient related risk factors or a single imaging modality would offer all aspects of needed staging information. The rationale for the present study is to find the most appropriate staging modality in high-risk PC at the time of initial staging.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed PC without previous PC treatment
* High-risk PC defined with one or more of the following criteria: Gleason ≥4+3, PSA ≥20, cT≥3a
* Adequate physical status defined (by treating clinician) as capability to undergo some form of active treatment for the PC and the physical status allowing the patient to undergo all study imaging modalities
* Signed informed consent

Exclusion Criteria:

* Previous PC treatment. Short-term androgen deprivation therapy is permitted if necessary for symptomatic and/or very high-risk PC patients
* Contraindications for MRI (cardiac pacemaker, intracranial clips etc.)
* Claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
To compare the diagnostic accuracy of 18F-PSMA-1007-PET/CT (PSMA-PET/CT) to 99mTc-HMDP planar bone scintigraphy (planar BS) in pessimistic, patient-based analysis detecting of bone metastases in the initial staging of high-risk PC patients. | 1 year
  Comparison of area under curve (AUC) values in receiver operating characteristic (ROC) curve of PSMA-PET/CT to planar BS in pessimistic, patient-based analysis detecting of bone metastases.
  The power calculations are made on the basis of previously published work, the SKELETA trial. To be able to detect the 0,19 difference (in AUC values) using a two-tailed test with a power of 80% at a significance level of 0.05 in a 2:1 ratio of sample sizes in negative/positive groups, 48 negative cases and 24 positive cases are required.
  Equivocal findings of the imaging modalities will be classified either as suggestive for metastases (pessimistic analysis) or suggestive for non-metastatic origin (optimistic analysis). AUC values will be calculated using the trapezoid rule and compared using a method described by Hanley and McNeil, two-sided p-values will be calculated.

SECONDARY OUTCOMES:
Sensitivity of each imaging modality will be measured in initial staging of nodal, soft tissue and bone metastasis | 1 year
  Sensitivity of PSMA-PET/CT, wbMRI, SPECT/CT, planar BS and wbCE-CT will be determined on patient-, regional- and lesion-level separately in detecting of nodal (regional lymph node/s), soft tissue (excluding regional nodal metastasis) and bone metastasis.
  The outcome measure unit is a percentage.
Specificity of each imaging modality will be measured in initial staging of nodal, soft tissue and bone metastasis | 1 year
  Specificity of PSMA-PET/CT, wbMRI, SPECT/CT, planar BS and wbCE-CT will be determined on patient-, regional- and lesion-level separately in detecting of nodal (regional lymph node/s), soft tissue (excluding regional nodal metastasis) and bone metastasis.
  The outcome measure unit is a percentage.
Diagnostic accuracy each imaging modality will be measured in initial staging of nodal, soft tissue and bone metastasis | 1 year
  Diagnostic accuracy of PSMA-PET/CT, wbMRI, SPECT/CT, planar BS and wbCE-CT will be determined on patient-, regional- and lesion-level separately in detecting of nodal (regional lymph node/s), soft tissue (excluding regional nodal metastasis) and bone metastasis.
  The outcome measure unit is a percentage.
The effect of staging on clinical treatment-decisions | 1 year
  The effect of staging on clinical treatment-decisions is based on clinical judgement done retrospectively by multi-disciplinary team consensus.
AUC values from receiver operating characteristic curve of each imaging modality will be measured in initial staging of nodal, soft tissue and bone metastasis | 1 year
  AUC values of PSMA-PET/CT, wbMRI, SPECT/CT, planar BS and wbCE-CT will be determined on patient-, regional- and lesion-level separately in detecting of nodal (regional lymph node/s), soft tissue (excluding regional nodal metastasis) and bone metastasis.
  The outcome measure is numeric unit 0-1.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, M.D.Ph.D, Principal Investigator — Department of urology, Turku University Hospital, VSSHP
Locations (1):
- Department of Urology, Turku, Finland

REFERENCES:
- [Background] Seikkula HA, Kaipia AJ, Rantanen ME, Pitkaniemi JM, Malila NK, Bostrom PJ. Stage-specific mortality and survival trends of prostate cancer patients in Finland before and after introduction of PSA. Acta Oncol. 2017 Jul;56(7):971-977. doi: 10.1080/0284186X.2017.1288298. Epub 2017 Feb 13. PMID 28406044
- [Background] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Background] Suh CH, Shinagare AB, Westenfield AM, Ramaiya NH, Van den Abbeele AD, Kim KW. Yield of bone scintigraphy for the detection of metastatic disease in treatment-naive prostate cancer: a systematic review and meta-analysis. Clin Radiol. 2018 Feb;73(2):158-167. doi: 10.1016/j.crad.2017.08.004. Epub 2017 Sep 25. PMID 28958581
- [Background] Even-Sapir E. Imaging of malignant bone involvement by morphologic, scintigraphic, and hybrid modalities. J Nucl Med. 2005 Aug;46(8):1356-67. PMID 16085595
- [Background] Van den Wyngaert T, Strobel K, Kampen WU, Kuwert T, van der Bruggen W, Mohan HK, Gnanasegaran G, Delgado-Bolton R, Weber WA, Beheshti M, Langsteger W, Giammarile F, Mottaghy FM, Paycha F; EANM Bone & Joint Committee and the Oncology Committee. The EANM practice guidelines for bone scintigraphy. Eur J Nucl Med Mol Imaging. 2016 Aug;43(9):1723-38. doi: 10.1007/s00259-016-3415-4. Epub 2016 Jun 4. PMID 27262701
- [Background] Even-Sapir E, Metser U, Mishani E, Lievshitz G, Lerman H, Leibovitch I. The detection of bone metastases in patients with high-risk prostate cancer: 99mTc-MDP Planar bone scintigraphy, single- and multi-field-of-view SPECT, 18F-fluoride PET, and 18F-fluoride PET/CT. J Nucl Med. 2006 Feb;47(2):287-97. PMID 16455635
- [Background] Helyar V, Mohan HK, Barwick T, Livieratos L, Gnanasegaran G, Clarke SE, Fogelman I. The added value of multislice SPECT/CT in patients with equivocal bony metastasis from carcinoma of the prostate. Eur J Nucl Med Mol Imaging. 2010 Apr;37(4):706-13. doi: 10.1007/s00259-009-1334-3. Epub 2009 Dec 17. PMID 20016889
- [Background] Silver DA, Pellicer I, Fair WR, Heston WD, Cordon-Cardo C. Prostate-specific membrane antigen expression in normal and malignant human tissues. Clin Cancer Res. 1997 Jan;3(1):81-5. PMID 9815541
- [Background] Eder M, Schafer M, Bauder-Wust U, Hull WE, Wangler C, Mier W, Haberkorn U, Eisenhut M. 68Ga-complex lipophilicity and the targeting property of a urea-based PSMA inhibitor for PET imaging. Bioconjug Chem. 2012 Apr 18;23(4):688-97. doi: 10.1021/bc200279b. Epub 2012 Mar 13. PMID 22369515
- [Background] Perera M, Papa N, Christidis D, Wetherell D, Hofman MS, Murphy DG, Bolton D, Lawrentschuk N. Sensitivity, Specificity, and Predictors of Positive 68Ga-Prostate-specific Membrane Antigen Positron Emission Tomography in Advanced Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Dec;70(6):926-937. doi: 10.1016/j.eururo.2016.06.021. Epub 2016 Jun 28. PMID 27363387
- [Background] Fendler WP, Schmidt DF, Wenter V, Thierfelder KM, Zach C, Stief C, Bartenstein P, Kirchner T, Gildehaus FJ, Gratzke C, Faber C. 68Ga-PSMA PET/CT Detects the Location and Extent of Primary Prostate Cancer. J Nucl Med. 2016 Nov;57(11):1720-1725. doi: 10.2967/jnumed.116.172627. Epub 2016 Jun 3. PMID 27261520
- [Background] Rhee H, Thomas P, Shepherd B, Gustafson S, Vela I, Russell PJ, Nelson C, Chung E, Wood G, Malone G, Wood S, Heathcote P. Prostate Specific Membrane Antigen Positron Emission Tomography May Improve the Diagnostic Accuracy of Multiparametric Magnetic Resonance Imaging in Localized Prostate Cancer. J Urol. 2016 Oct;196(4):1261-7. doi: 10.1016/j.juro.2016.02.3000. Epub 2016 May 21. PMID 27220897
- [Background] van Leeuwen PJ, Emmett L, Ho B, Delprado W, Ting F, Nguyen Q, Stricker PD. Prospective evaluation of 68Gallium-prostate-specific membrane antigen positron emission tomography/computed tomography for preoperative lymph node staging in prostate cancer. BJU Int. 2017 Feb;119(2):209-215. doi: 10.1111/bju.13540. Epub 2016 Jun 18. PMID 27207581
- [Background] Janssen JC, Meissner S, Woythal N, Prasad V, Brenner W, Diederichs G, Hamm B, Makowski MR. Comparison of hybrid 68Ga-PSMA-PET/CT and 99mTc-DPD-SPECT/CT for the detection of bone metastases in prostate cancer patients: Additional value of morphologic information from low dose CT. Eur Radiol. 2018 Feb;28(2):610-619. doi: 10.1007/s00330-017-4994-6. Epub 2017 Aug 4. PMID 28779400
- [Background] Cardinale J, Schafer M, Benesova M, Bauder-Wust U, Leotta K, Eder M, Neels OC, Haberkorn U, Giesel FL, Kopka K. Preclinical Evaluation of 18F-PSMA-1007, a New Prostate-Specific Membrane Antigen Ligand for Prostate Cancer Imaging. J Nucl Med. 2017 Mar;58(3):425-431. doi: 10.2967/jnumed.116.181768. Epub 2016 Oct 27. PMID 27789722
- [Background] Kesch C, Vinsensia M, Radtke JP, Schlemmer HP, Heller M, Ellert E, Holland-Letz T, Duensing S, Grabe N, Afshar-Oromieh A, Wieczorek K, Schafer M, Neels OC, Cardinale J, Kratochwil C, Hohenfellner M, Kopka K, Haberkorn U, Hadaschik BA, Giesel FL. Intraindividual Comparison of 18F-PSMA-1007 PET/CT, Multiparametric MRI, and Radical Prostatectomy Specimens in Patients with Primary Prostate Cancer: A Retrospective, Proof-of-Concept Study. J Nucl Med. 2017 Nov;58(11):1805-1810. doi: 10.2967/jnumed.116.189233. Epub 2017 May 4. PMID 28473595
- [Background] Freitag MT, Kesch C, Cardinale J, Flechsig P, Floca R, Eiber M, Bonekamp D, Radtke JP, Kratochwil C, Kopka K, Hohenfellner M, Stenzinger A, Schlemmer HP, Haberkorn U, Giesel F. Simultaneous whole-body 18F-PSMA-1007-PET/MRI with integrated high-resolution multiparametric imaging of the prostatic fossa for comprehensive oncological staging of patients with prostate cancer: a pilot study. Eur J Nucl Med Mol Imaging. 2018 Mar;45(3):340-347. doi: 10.1007/s00259-017-3854-6. Epub 2017 Oct 16. PMID 29038888
- [Background] Backhaus P, Noto B, Avramovic N, Grubert LS, Huss S, Bogemann M, Stegger L, Weckesser M, Schafers M, Rahbar K. Targeting PSMA by radioligands in non-prostate disease-current status and future perspectives. Eur J Nucl Med Mol Imaging. 2018 May;45(5):860-877. doi: 10.1007/s00259-017-3922-y. Epub 2018 Jan 15. PMID 29335762
- [Background] Venkitaraman R, Cook GJ, Dearnaley DP, Parker CC, Khoo V, Eeles R, Huddart RA, Horwich A, Sohaib SA. Whole-body magnetic resonance imaging in the detection of skeletal metastases in patients with prostate cancer. J Med Imaging Radiat Oncol. 2009 Jun;53(3):241-7. doi: 10.1111/j.1754-9485.2009.02070.x. PMID 19624290
- [Background] Lecouvet FE, Geukens D, Stainier A, Jamar F, Jamart J, d'Othee BJ, Therasse P, Vande Berg B, Tombal B. Magnetic resonance imaging of the axial skeleton for detecting bone metastases in patients with high-risk prostate cancer: diagnostic and cost-effectiveness and comparison with current detection strategies. J Clin Oncol. 2007 Aug 1;25(22):3281-7. doi: 10.1200/JCO.2006.09.2940. PMID 17664475
- [Background] Pasoglou V, Michoux N, Peeters F, Larbi A, Tombal B, Selleslagh T, Omoumi P, Vande Berg BC, Lecouvet FE. Whole-body 3D T1-weighted MR imaging in patients with prostate cancer: feasibility and evaluation in screening for metastatic disease. Radiology. 2015 Apr;275(1):155-66. doi: 10.1148/radiol.14141242. Epub 2014 Dec 15. PMID 25513855
- [Background] Hovels AM, Heesakkers RA, Adang EM, Jager GJ, Strum S, Hoogeveen YL, Severens JL, Barentsz JO. The diagnostic accuracy of CT and MRI in the staging of pelvic lymph nodes in patients with prostate cancer: a meta-analysis. Clin Radiol. 2008 Apr;63(4):387-95. doi: 10.1016/j.crad.2007.05.022. Epub 2008 Feb 4. PMID 18325358
- [Background] Thoeny HC, Froehlich JM, Triantafyllou M, Huesler J, Bains LJ, Vermathen P, Fleischmann A, Studer UE. Metastases in normal-sized pelvic lymph nodes: detection with diffusion-weighted MR imaging. Radiology. 2014 Oct;273(1):125-35. doi: 10.1148/radiol.14132921. Epub 2014 Jun 2. PMID 24893049
- [Background] Jambor I, Kuisma A, Ramadan S, Huovinen R, Sandell M, Kajander S, Kemppainen J, Kauppila E, Auren J, Merisaari H, Saunavaara J, Noponen T, Minn H, Aronen HJ, Seppanen M. Prospective evaluation of planar bone scintigraphy, SPECT, SPECT/CT, 18F-NaF PET/CT and whole body 1.5T MRI, including DWI, for the detection of bone metastases in high risk breast and prostate cancer patients: SKELETA clinical trial. Acta Oncol. 2016;55(1):59-67. doi: 10.3109/0284186X.2015.1027411. Epub 2015 Apr 2. PMID 25833330
- [Background] Cardinale J, Martin R, Remde Y, Schafer M, Hienzsch A, Hubner S, Zerges AM, Marx H, Hesse R, Weber K, Smits R, Hoepping A, Muller M, Neels OC, Kopka K. Procedures for the GMP-Compliant Production and Quality Control of [18F]PSMA-1007: A Next Generation Radiofluorinated Tracer for the Detection of Prostate Cancer. Pharmaceuticals (Basel). 2017 Sep 27;10(4):77. doi: 10.3390/ph10040077. PMID 28953234
- [Background] Trajman A, Luiz RR. McNemar chi2 test revisited: comparing sensitivity and specificity of diagnostic examinations. Scand J Clin Lab Invest. 2008;68(1):77-80. doi: 10.1080/00365510701666031. PMID 18224558
- [Background] Hanley JA, McNeil BJ. A method of comparing the areas under receiver operating characteristic curves derived from the same cases. Radiology. 1983 Sep;148(3):839-43. doi: 10.1148/radiology.148.3.6878708.
- [Background] Even-Sapir E, Metser U, Flusser G, Zuriel L, Kollender Y, Lerman H, Lievshitz G, Ron I, Mishani E. Assessment of malignant skeletal disease: initial experience with 18F-fluoride PET/CT and comparison between 18F-fluoride PET and 18F-fluoride PET/CT. J Nucl Med. 2004 Feb;45(2):272-8. PMID 14960647
- [Background] Lecouvet FE, El Mouedden J, Collette L, Coche E, Danse E, Jamar F, Machiels JP, Vande Berg B, Omoumi P, Tombal B. Can whole-body magnetic resonance imaging with diffusion-weighted imaging replace Tc 99m bone scanning and computed tomography for single-step detection of metastases in patients with high-risk prostate cancer? Eur Urol. 2012 Jul;62(1):68-75. doi: 10.1016/j.eururo.2012.02.020. Epub 2012 Feb 17. PMID 22366187
- [Background] Vanel D, Bittoun J, Tardivon A. MRI of bone metastases. Eur Radiol. 1998;8(8):1345-51. doi: 10.1007/s003300050549. PMID 9853211
- [Background] Schmidt GP, Schoenberg SO, Schmid R, Stahl R, Tiling R, Becker CR, Reiser MF, Baur-Melnyk A. Screening for bone metastases: whole-body MRI using a 32-channel system versus dual-modality PET-CT. Eur Radiol. 2007 Apr;17(4):939-49. doi: 10.1007/s00330-006-0361-8. Epub 2006 Sep 2. PMID 16951929
- [Derived] Kivikallio A, Malaspina S, Saarinen I, Seppanen M, Anttinen M, Jambor I, Verho J, Kemppainen J, Aronen HJ, Bostrom PJ, Ettala O, Taimen P. Prospective comparison of 18F-PSMA-1007 PET/CT and MRI with histopathology as the reference standard for intraprostatic tumour detection and T-staging of high-risk prostate cancer. Eur J Nucl Med Mol Imaging. 2025 Aug;52(10):3709-3719. doi: 10.1007/s00259-025-07208-z. Epub 2025 Mar 31. PMID 40159542
- [Derived] Malaspina S, Anttinen M, Taimen P, Jambor I, Sandell M, Rinta-Kiikka I, Kajander S, Schildt J, Saukko E, Noponen T, Saunavaara J, Dean PB, Sequeiros RB, Aronen HJ, Kemppainen J, Seppanen M, Bostrom PJ, Ettala O. Prospective comparison of 18F-PSMA-1007 PET/CT, whole-body MRI and CT in primary nodal staging of unfavourable intermediate- and high-risk prostate cancer. Eur J Nucl Med Mol Imaging. 2021 Aug;48(9):2951-2959. doi: 10.1007/s00259-021-05296-1. Epub 2021 Mar 13. PMID 33715033
- [Derived] Anttinen M, Ettala O, Malaspina S, Jambor I, Sandell M, Kajander S, Rinta-Kiikka I, Schildt J, Saukko E, Rautio P, Timonen KL, Matikainen T, Noponen T, Saunavaara J, Loyttyniemi E, Taimen P, Kemppainen J, Dean PB, Blanco Sequeiros R, Aronen HJ, Seppanen M, Bostrom PJ. A Prospective Comparison of 18F-prostate-specific Membrane Antigen-1007 Positron Emission Tomography Computed Tomography, Whole-body 1.5 T Magnetic Resonance Imaging with Diffusion-weighted Imaging, and Single-photon Emission Computed Tomography/Computed Tomography with Traditional Imaging in Primary Distant Metastasis Staging of Prostate Cancer (PROSTAGE). Eur Urol Oncol. 2021 Aug;4(4):635-644. doi: 10.1016/j.euo.2020.06.012. Epub 2020 Jul 13. PMID 32675047